CLINICAL TRIAL: NCT05943587
Title: The Development and Evaluation of Culturally Sensitive Pain Neuroscience Education in Children With Chronic Pain
Brief Title: The Development and Evaluation of Pain Neuroscience Education in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-127
Record Dates: First submitted 2023-05-31; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain; Child, Only
Keywords: Chronic Pain; Children; Pain Neuroscience Education; Physical Therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, Modified Delphi Study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic pain group (Experimental): 30-45 minute individual sessions of culture-sensitive PNE4kids training will be applied.
  Interventions: Other: culture-sensitive PNE4kids
- Control Group (Active Comparator): 30-45 minute individual sessions of standard education training will be applied.
  Interventions: Other: standard education

INTERVENTIONS:
Other: culture-sensitive PNE4kids — Culturally adapted PNE4kids used by physiotherapists worldwide in chronic pain rehabilitation.
  Arms: Chronic pain group
Other: standard education — Standard education used by physiotherapists worldwide in chronic pain rehabilitation.
  Arms: Control Group

SUMMARY:
The International Association for the Study of Pain and The International Classification of Diseases (ICD) 11 define chronic pain as pain lasting more than 3 months, regardless of the cause. For children and adolescents, chronic pain is an extremely terrible and suffering problem. Periods of persistent pain negatively affect the child's participation in school and recreational activities, leading to academic problems and social exclusion. Moreover, children are at increased risk of experiencing chronic pain problems in adulthood. Because of these difficulties children with chronic pain should be treated as soon as possible. Pain Neuroscience Education (PNE) is an educational approach used in chronic pain rehabilitation. The purpose of PNE is to change individual's perception of pain. The most fundamental and crucial aspect of PNE is educating patients about the underlying causes of their pain. The primary purpose of the project is to conduct a modified Delphi survey to obtain and synthesize expert opinions on PNE materials. The second aim of this study is to investigate the effect of PNE on pain, quality of life and participation in children with chronic pain and compare it with the standard treatment program.

DETAILED DESCRIPTION:
Chronic pain is not directly cause death but it is a major source of disability and suffering. Because of the enormous medical, economic, and social burden of chronic pain worldwide better understanding of pain biology has become a critical topic in order to develop targeted, novel, safe, and effective treatments. Pain Neuroscience Education (PNE) is a multidisciplinary educational method used by physiotherapists worldwide in chronic pain rehabilitation. The goal of PNE is to alter a person's perception of pain. PNE aims to correct patient misconceptions about pain physiology. As a result, pain education can help to reduce levels of fear of pain, fear of movement, pain catastrophizing thoughts, and passive coping strategies (for example, the use of painkillers or massage treatments). Currently, only a few research have investigated the benefits of PNE in children. The majority of studies have focused on pain management education programs rather than explaining the neurology of pain. The combined effects of PNE and physiotherapy have not been studied in children. But adult studies are demonstrated that PNE and physiotherapy are effective. According to studies, PNE has been linked to promising results in the treatment of chronic pain and functional impairment in adults. James et al. concluded that PNE reduced pain, disability, pain catastrophization, and kinesiophobia in the short and medium term, based on a systematic evaluation of 12 randomized controlled studies assessing the effect of PNE in individuals with chronic musculoskeletal pain. Currently, no study has been conducted in investigators country that has adapted PNE for children and evaluated the consequences of PNE use. The primary aim of the research is to perform a modified Delphi survey to obtain and synthesize expert opinions on culturally appropriate PNE materials for children in terms of content, relevance of information, clarity and intelligibility of information, and visual qualities of the materials. The second aim of the research is to investigate the impacts of culturally tailored PNE on pain symptoms (pain severity, pain awareness, fear of pain, catastrophizing pain, dealing with pain), quality of life, and involvement in children with chronic pain, as well as to compare it to a normal education program.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 years and 12 years;
* Diagnosed with chronic pain (at least three months of pain and a pain frequency of three or more days per week)
* Those who do not take analgesics 48 hours prior to study evaluations.

Exclusion Criteria:

* Patients with unmanageable psychological disorders (e.g., attention deficit hyperactivity disorder, autistic spectrum disorder, schizophrenia, bipolar disorder, major depressive disorder) would be excluded from the study.

Patients who started a new treatment during the trial or 6 weeks before to the study for chronic pain.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Scale | change from baseline to end of the 1 week and 4 weeks
  It is a valid and reliable scale preferred by children and their families to evaluate the severity of pain. It consists of 6 facial expressions that symbolize the severity of pain. These show the stages of increased pain from a smiling face (0 points) to a very sad and crying face (10 points). The meaning of each facial expression is carefully explained to the child. Children rate pain intensity according to face shapes.It consists of 6 facial expressions that symbolize the severity of the pain. It is scored between 0-10. Increasing scores indicate more pain.
Pain Vigilance and Awareness Questionnaire Child & Adult Version | change from baseline to end of the 1 week and 4 weeks
  Pain Vigilance and Awareness Questionnaire Child evaluates children's attention to pain. There are 14 items on the scale. A 0-5 likert scale is used for scoring. It has a rating of 0 (never) to 5 (always) (always). The total score is calculated by multiplying the individual item scores. Pain Vigilance and Awareness Questionnaire-Adult uses 16 items to test adults' attention and pain awareness. It has ten items for paying attention and six ones for being aware. A 0-5 likert scale is used for scoring. 0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = almost always, and 5 = always. The scale's eighth and sixteenth items are scored in reverse order. The scaled total score ranges from 0 to 80. Higher ratings suggest that you are more conscious of your pain.Items are rated on a 6-point scale, ranging from 0 (never) to 5 (always). The 8th and 16th items of the scale are reverse scored. The scale total score is obtained between 0-80. Higher scores indicate greater awareness of pain.
Fear of Pain Questionnaire for Children/Parents | change from baseline to end of the 1 week and 4 weeks
  The Fear of Pain Questionnaire for Children-Short Form is a 10-item version of the 24-item Fear of Pain Questionnaire for Children. It uses children's self-reports to assess pain-related fears (4 items) and avoidance behaviours (6 items). A 0-4 Likert scale is used for scoring. A score of 0 indicates strong disagreement, while a score of 5 indicates strong agreement.Items are summed to derive a total score (with between 0-40) . Higher scores indicate higher pain-related fear and avoidance behaviors.
Pain Catastrophizing Scale- Child | change from baseline to end of the 1 week and 4 weeks
  Crombez et al. created the Pain Catastrophizing Scale-Child, an adaptation of the Pain Catastrophizing Scale for children. Catastrophizing behaviours is evaluated with 13 items: rumination (4 items), magnification (3 items), and helplessness (6 items). The scoring is done on a 0-4 point Likert scale. It is evaluated on a scale of 0 (not at all) to 4 (very extremely).Items are summed to derive a total score (with between 0-52), with higher scores indicating more pain catastrophizing.
Functional Disability Inventory | change from baseline to end of the 1 week and 4 weeks
  Walker and Greene developed the Functional Disability Inventory to assess challenges faced by school-age children and adolescents in executing activities of daily living from the child's perspective. There are 15 items in Functional Disability Inventory. Each item asks about how many physical challenges or obstacles the youngster has experienced while executing the activity in the previous few days. The scoring is done on a 0-4 point Likert scale. It is ranked between 0 (no problem) and 4 (impossible). Items are summed to derive a total score (with between 0-60) , with higher total scores indicating greater disability.
Pain Coping Questionnaire | change from baseline to end of the 1 week and 4 weeks
  Evaluates the coping strategies of children and adolescents with a total of 39 items in 8 subscales. These are seeking knowledge, problem solving, seeking social support, positive self-suggestion, behavioural distraction, cognitive distraction, externalization, and internalization/catastrophizing. Items are assessed on a 5-point Likert scale, with 1 indicating never and 5 indicating very often. Higher ratings indicate higher use of coping strategy. PCQ consists of parent and adolescent form.The scores for each subscale are calculated by averaging the items. Higher scores indicate that the child uses strategies to cope more frequently.

SECONDARY OUTCOMES:
Participation and Environment- Children and Youth | change from baseline to end of the 1 week and 4 weeks
  The participation sections included 10 activities in the home setting, five activities in the school setting, and 10 in the community setting. For each activity, the range of participation is daily to never, with scores between 0 and 8; higher scores indicate greater participation. The range of involvement is from very involved to minimally involved, with scores between 1 and 5; higher scores indicate greater involvement. The range of whether change is desired in the child's participation in this kind of activity is no or yes, with scores between 0 and 1. Environmental features supports and barriers (e.g., do the features of the environment help or make it harder?) for the child to participate in activities at home, school, or in a community setting with scores between 1 and 4; increased scores indicate environmental help.
Pediatric Quality of Life Inventory | change from baseline to end of the 1 week and 4 weeks
  Pediatric Quality of Life Inventory is a health-related quality-of-life scale for children and adolescents aged 2 to 18. There are three areas in which you can score. The first is the scale total score, followed by the physical health total score, and finally the psychosocial health total score, which is calculated from the item scores assessing emotional, social, and school functions. The Pediatric Quality of Life Inventory is a 23-item quality of life scale that is appropriate for use in large groups such as schools and hospitals, as well as in both healthy and unhealthy children and adolescents. The items are graded on a scale of 0 to 100. The answer is scored 100 if it is marked as never, 75 if it is marked as rarely, 50 if it is marked as occasionally, 25 if it is marked as frequently, and 0 if it is marked as almost constantly. The higher the total PedsQL score, the higher the perceived health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Assoc. Prof., Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracey I, Mantyh PW. The cerebral signature for pain perception and its modulation. Neuron. 2007 Aug 2;55(3):377-91. doi: 10.1016/j.neuron.2007.07.012. PMID 17678852
- [Background] Pas R, Meeus M, Malfliet A, Baert I, Oosterwijck SV, Leysen L, Nijs J, Ickmans K. Development and feasibility testing of a Pain Neuroscience Education program for children with chronic pain: treatment protocol. Braz J Phys Ther. 2018 May-Jun;22(3):248-253. doi: 10.1016/j.bjpt.2018.02.004. Epub 2018 Mar 4. PMID 29550259
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Malfliet A, Leysen L, Pas R, Kuppens K, Nijs J, Van Wilgen P, Huysmans E, Goudman L, Ickmans K. Modern pain neuroscience in clinical practice: applied to post-cancer, paediatric and sports-related pain. Braz J Phys Ther. 2017 Jul-Aug;21(4):225-232. doi: 10.1016/j.bjpt.2017.05.009. Epub 2017 May 19. PMID 28579013
- [Background] Nijs J, Torres-Cueco R, van Wilgen CP, Girbes EL, Struyf F, Roussel N, van Oosterwijck J, Daenen L, Kuppens K, Vanwerweeen L, Hermans L, Beckwee D, Voogt L, Clark J, Moloney N, Meeus M. Applying modern pain neuroscience in clinical practice: criteria for the classification of central sensitization pain. Pain Physician. 2014 Sep-Oct;17(5):447-57. PMID 25247901
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Robins H, Perron V, Heathcote LC, Simons LE. Pain Neuroscience Education: State of the Art and Application in Pediatrics. Children (Basel). 2016 Dec 21;3(4):43. doi: 10.3390/children3040043. PMID 28009822
- [Background] Siddall B, Ram A, Jones MD, Booth J, Perriman D, Summers SJ. Short-term impact of combining pain neuroscience education with exercise for chronic musculoskeletal pain: a systematic review and meta-analysis. Pain. 2022 Jan 1;163(1):e20-e30. doi: 10.1097/j.pain.0000000000002308. PMID 33863860